CLINICAL TRIAL: NCT01632696
Title: Open-label, Single Arm, Tumor Imaging and Dosimetry Study of I-124 PGN650 in Advanced Solid Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PPHM 1201
Record Dates: First submitted 2012-06-12; First posted 2012-07-03 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Malignant Solid Tumor
Keywords: Antibodies, Monoclonal; Biologics; F(ab')2; Positron-emission tomography (PET); Phosphatidylserine (PS); Solid Tumors; Tumor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-124 PGN650 for PET/CT (Experimental)
  Interventions: Drug: I-124 PGN650 for PET/CT

INTERVENTIONS:
Drug: I-124 PGN650 for PET/CT — I-124 PGN650 for PET/CT Day 1, Day 2 and 3.
  Other Names: I-124 PGN650

SUMMARY:
Tumor Imaging of I-124 PGN65 in Solid Tumors

DETAILED DESCRIPTION:
Up to 12 patients (6 men and 6 women) will be enrolled in this open-label, single-arm, tumor imaging and dosimetry study of I-124 PGN650 in solid tumors. All eligible patients who give written, informed consent and meet all inclusion criteria and no exclusion criteria, and whose laboratory results are within specified limits at the screening visit, will be enrolled. All study subjects will receive a single intravenous (IV) dose of I-124 PGN650. Study subjects will have whole body PET/CT imaging at three different timepoints with all patients having PET/CT at 0 to 60 minutes after injection of I-124 PGN650. Study subjects will then be assigned to either a 3 to 5-hour or 6 to 8-hour timepoint and either an 18 to 26 hour or 42 to 52 hour post-injection timepoint. Tumor and whole body radioactivity distribution will be measured.

ELIGIBILITY:
Inclusion Criteria

1. Signed informed consent form.
2. Male or female, ≥ 18 years of age.
3. Histologically or cytologically confirmed solid tumors at any stage with at least one lesion (primary, metastatic, or recurrent) ≥ 1.5 cm in diameter documented by CT. If the lesion is located in a lymph node, the shortest diameter of the lymph node must be ≥ 1.5 cm as defined by RECIST 1.1. (Note: See Exclusion Criteria #1.)
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Adequate baseline hematological and organ function, assessed by laboratory values prior to study treatment as follows: absolute neutrophil count (ANC) > 1.0 x 109/L; hemoglobin > 7 g/dL; serum creatinine < 2 x institutional upper limit of normal (IULN); aspartate transaminase (AST) < 2.5 x IULN; alanine transaminase (ALT) < 2.5 x IULN; (if liver metastases are present, ALT and AST < 5 x IULN); total bilirubin < 1.5 x IULN.
6. Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence), for the duration of study participation (i.e., from dosing day 1 until study day 8). Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
7. Patient must be willing and able to undergo the imaging studies outlined in the protocol.

Exclusion Criteria

1. Only measureable disease (primary or metastatic) is located in or near the thyroid gland, liver, kidney, or urinary bladder.
2. Medical conditions such as ischemic heart or lung disease that may be considered an unacceptable risk.
3. Females who are lactating or pregnant.
4. Persistent acute toxicities from prior anti-cancer therapy.
5. History of hypersensitivity to iodine.
6. Known bladder outlet obstruction.
7. Any condition that would in the Investigator's judgment prevents compliance with the requirements of the protocol.
8. Patients with known history of an autoimmune disease- including but not limited to: celiac disease, Crohn's disease, dermatomyositis, Grave's disease, systemic lupus erythematosus, myasthenia gravis, psoriasis, and rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
To estimate the intensity and distribution in critical and non-critical organs. | Day 1
To estimate the intensity and distribution in critical and non-critical organs. | Day 2
To estimate the intensity and distribution in critical and non-critical organs. | Day 3

SECONDARY OUTCOMES:
The presence of tumor imaging using I-124 PGN650 as a PS-targeting agent. | Day 1, Day 2 and Day 3
Demonstrate the safety of tumor imaging in patients with solid cancers. | Day 1, Day 2 and Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehsashti, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri, United States